CLINICAL TRIAL: NCT03084809
Title: Clinical Efficacy of Chemotherapy Combined With Cytokine-induced Killer in Treatment of Patients With Colon Cancer
Brief Title: Chemotherapy Combined With CIK Treating Colon Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China Meitan General Hospital (Other)
Responsible Party: Principal Investigator, Hao Peng, Principal investigator, China Meitan General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIK-2
Record Dates: First submitted 2017-03-08; First posted 2017-03-21 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Colorectal Cancer; Cytokine-induced Killer Cells; Postoperative Complications; Survival
MeSH Terms: conditions — Colorectal Neoplasms; Postoperative Complications | interventions — Oxaliplatin; Leucovorin; Fluorouracil; Folfox protocol

STUDY DESIGN:
Intervention Model Description: Group 1: chemotherapy (5-Fluorouridine, leucovorin and oxaliplatin [FOLFOX4]) combined with cytokine-induced killer cells (CIK) Group 2: chemotherapy (5-Fluorouridine, leucovorin and oxaliplatin [FOLFOX4])
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cytokine-induced killer cells + FOLFOX4 (Experimental): Cytokine-induced killer cells + FOLFOX4 intervention:
  Day 1: Oxaliplatin 130 mg/m² IV infusion in 500 mL 5% dextrose in water (D5W); Day 2-6: leucovorin 200mg/m² IV infusion in D5W both given over 2 hours at the same time in separate bags; Day 2-6: 5-FU 500 mg/m² IV bolus given continuously over 4-6 hours.The treatment is given for 4-6 cycles, every 3 weeks.
  Collected cytokine-induced killer cells (CIK) cells were suspended with 100ml saline (containing 5ml 20% human serum albumin) and given continuously over 2 hours/ day for 3 days.
  Interventions: Drug: Cytokine-induced killer cells+ FOLFOX4
- FOLFOX4 (Experimental): FOLFOX4 intervention:
  Day 1: Oxaliplatin 130 mg/m² IV infusion in 500 mL 5% dextrose in water (D5W); Day 2-6: leucovorin 200mg/m² IV infusion in D5W both given over 2 hours at the same time in separate bags; Day 2-6: 5-FU 500 mg/m² IV bolus given continuously over 4-6 hours. The treatment is given for 4-6 cycles, every 3 weeks.
  Interventions: Drug: FOLFOX4

INTERVENTIONS:
Drug: Cytokine-induced killer cells+ FOLFOX4 — Day 1: Oxaliplatin 130 mg/m² IV infusion in 500 mL D5W. Day 2-6: leucovorin 200mg/m² IV infusion in D5W both given over 2 hours at the same time in separate bags Day 2-6: 5-FU 500 mg/m² IV bolus given continuously over 4-6 hours. The treatment is given for 4-6 cycles, every 3 weeks. Collected CIK cells were suspended with 100ml saline (containing 5ml 20% human serum albumin) and given continuously over 2 hours/ day for 3 days.
  Other Names: CIK + Oxaliplatin + leucovorin + 5-FU
  Arms: Cytokine-induced killer cells + FOLFOX4
Drug: FOLFOX4 — Day 1: Oxaliplatin 130 mg/m² IV infusion in 500 mL D5W. Day 2-6: leucovorin 200mg/m² IV infusion in D5W both given over 2 hours at the same time in separate bags Day 2-6: 5-FU 500 mg/m² IV bolus given continuously over 4-6 hours. The treatment is given for 4-6 cycles, every 3 weeks.
  Other Names: Oxaliplatin + leucovorin + 5-FU
  Arms: FOLFOX4

SUMMARY:
Cytokine-induced killer cells (CIK) is an auxiliary antitumor treatment. The investigators aim to evaluate the clinical efficacy of chemotherapy combined with CIK in the treatment of postoperative colorectal cancer patients. And to provide useful reference for the clinical application of CIK in colorectal cancer patients.

DETAILED DESCRIPTION:
Over the past decade, advances in combination chemotherapy regimens for colorectal cancer have led to significant improvement in progression-free and overall survival. Cytokine-induced killer cells (CIK) is an auxiliary antitumor treatment. Research has demonstrated the median overall survival (OS) in patients received CIK combined with chemotherapy (5-Fluorouridine, leucovorin and oxaliplatin [FOLFOX4] plan) was significantly increased compared with that in patients received chemotherapy alone. Furthermore, there was a trend toward superior progression-free survival time (PFS) in patients received CIK combined with chemotherapy compared with that in patients received chemotherapy alone. The investigators aim to evaluate the clinical efficacy of chemotherapy (FOLFOX4) combined with CIK in the treatment of postoperative colorectal cancer patients. And to provide useful reference for the clinical application of CIK in colorectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Tumor, Nodes, Metastasis (TNM) stage of II or III;
2. Patients received radical resection of colon cancer;
3. Pathological diagnosis of adenocarcinoma;
4. Patients not received radiotherapy and chemotherapy before surgery;
5. The preoperative examination confirmed without systemic metastasis;
6. Patient has the Karnofsky score more than 70 points;
7. Subjects signed informed consent.

Exclusion Criteria:

1. Patients who was serious allergy to any of the ingredients of drugs used in this study;
2. Patients who unable to comply with the treatment plan or research program;
3. Patients with severe systemic disease that the researchers judged will be unable to complete the study;
4. Patients have severe heart disease, such as myocardial infarction within 6 months;
5. Patients who have received chemotherapy or systemic antitumor therapy (such as monoclonal antibody therapy);
6. Patients received radiotherapy;
7. Having other malignant tumors in the last 5 years, but not including who has been cured through surgery and survived 5 year of disease-free;
8. Any unstable systemic diseases (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, or myocardial infarction, serious arrhythmias, liver, kidney or metabolic diseases within six months).
9. Patients who do not get effective treatment of inflammation, eye infections or predisposing factors;
10. Physical examination or laboratory findings evidence reasonable doubt who is ill or use of related drugs could affect the study;
11. Patients with serious active infections;
12. Woman who are pregnant or lactating.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-05-06 (Actual); Primary Completion 2014-09-15 (Actual); Study Completion 2014-09-15 (Actual)

PRIMARY OUTCOMES:
Relapse Free Survival in 2 years | 2 years (24 months)

SECONDARY OUTCOMES:
Relapse Free Survival in 3 years | Follow-up: 3 years
5 year Overall Survival | Follow-up: 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Li-Min Wang, Dr., Principal Investigator — Center for Drug Evaluation, China food and Drug Administration

IPD SHARING:
Plan to Share IPD: Undecided
whether individual participant data (IPD) could be shared must obtain the consent of the subjects